CLINICAL TRIAL: NCT04706871
Title: Transcutaneous Auricular Vagus Nerve Stimulation in the Treatment of Functional Dyspepsia : A Randomized Controlled Trial
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation Treatment on Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: taVNS-FD-2018
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Functional Dyspepsia
Keywords: transcutaneous auricular vagus nerve stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS group (Experimental)
  Interventions: Device: taVNS
- tnVNS group (Placebo Comparator)
  Interventions: Device: tnVNS

INTERVENTIONS:
Device: taVNS — taVNS was applied using a Huatuo stimulator (SDZ-IIB) developed by Suzhou manufacture of Medical Device and Material. Stimulation parameters was 1 mA of electrical current at a frequency of 30 Hz with pulse duration ≤ 1 ms, for 30min, administered twice daily.
  The two electrodes were placed on the cymba conchae and concha around the left ear.
  Arms: taVNS group
Device: tnVNS — tnVNS was applied using a Huatuo stimulator (SDZ-IIB) developed by Suzhou manufacture of Medical Device and Material. Stimulation parameters was 1 mA of electrical current at a frequency of 30 Hz with pulse duration ≤ 1 ms, for 30min, administered twice daily.
  The two electrodes were placed on the antihelix around the left ear.
  Arms: tnVNS group

SUMMARY:
Objective: To observe the effect of the treatment of transcutaneous auricular vagus nerve stimulation (taVNS) for the functional dyspepsia (FD).

Methods: We accrued 94 patients at Beijing TongRen Hospital. All treatments were self-administered by the patients at home after training at the hospital. Patients completed questionnaires at baseline and after 4 weeks, 8 weeks, 12 weeks. The FD Symptoms Index, Functional Dyspepsia Quality of Life Scale (FDDQL), Hamilton Anxiety Scale (HAMA), Hamilton Depression Scale (HAMD), and Self-Depression Rating Scale (SDS) were performed to evaluate the therapeutic effects.

A difference of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age >=18 and Age <=65. 2. Clinical diagnosis of functional dyspepsia.

Exclusion Criteria:

* 1. History of depression, tumors, thyroid disease, diabetes, cardiac diseases. 2. History of gastrointestinal surgery. 3. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline in the FD Symptoms Index at 16 Weeks | Day 0, 4-weeks, postintervention at Week 4, postintervention at Week 12
  FD Symptoms Index to measure the subjective symptoms of dyspepsia.
Mean change from Baseline in the FDQOL at 16 Weeks | Day 0, 4-weeks, postintervention at Week 4, postintervention at Week 12
  FDQOL to measure the subjective quality of life.

SECONDARY OUTCOMES:
Mean change from Baseline in the HAMA at 16 Weeks | Day 0, 4-weeks, postintervention at Week 4, postintervention at Week 12
  HAMA to measure the subjective anxiety symptoms
Mean change from Baseline in the HAMD at 16 Weeks | Day 0, 4-weeks, postintervention at Week 4, postintervention at Week 12
  HAMD to measure the subjective depression symptoms
Mean change from Baseline in the SDS at 16 Weeks | Day 0, 4-weeks, postintervention at Week 4, postintervention at Week 12
  SDS to measure the subjective depression symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No